CLINICAL TRIAL: NCT03040128
Title: Minocycline and Matrix Metalloproteinase Inhibition in Acute Intracerebral Hemorrhage: A Pilot Trial
Brief Title: Use of Minocycline in Intracerebral Hemorrhage
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Principal Investigator, Jason Chang, Principal Investigator, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MITCH
Record Dates: First submitted 2017-01-25; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: random number generator (placebo vs. study drug)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): normal saline infusion
  Interventions: Other: normal saline infusion
- minocycline (Experimental): intravenous minocycline
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — high-dose, intravenous minocycline
  Arms: minocycline
Other: normal saline infusion
  Arms: placebo

SUMMARY:
To date, no neuroprotective drugs have demonstrated clinical efficacy in intracerebral hemorrhage (ICH). This study will use intravenous (IV) minocycline in ICH to evaluate for (1) safety/ tolerability and (2) evaluate for clinical efficacy

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) remains a devastating neurological disorder with high mortality and poor prognosis with unchanged mortality rates (53-59%). Acute treatment options for ICH remain supportive with no available effective drug or surgical therapy. All trials so far have failed to improve clinical outcome in randomized, double-blinded trials. However, one area of interest has been maintaining the integrity of the blood-brain-barrier (BBB) and preventing the growth of vasogenic edema. Matrix metalloproteinases (MMP) are a family of ubiquitous zinc-dependent endopeptidase enzymes whose primary function is the digestion of collagen type IV, laminin, and fibronectin for the purpose of remodeling extracellular basal lamina. Elevated MMP-9 as a pathological process associated with larger hematoma volume, larger perihematomal edema, and poorer clinical outcome in intracerebral hemorrhage is well documented in animal models and patients. One particular MMP-9 inhibitor gaining usage in cerebrovascular disease is minocycline. Normally FDA-approved for bacterial infection and acne vulgaris, minocycline has also been found to be both a safe and effective treatment in ischemic stroke; its potential role as a neuroprotectant in ischemic stroke is currently being tested in a large, randomized, double-blinded trial. Minocycline's beneficial role as a neuroprotectant may also extend to ICH. By inhibiting MMP-9, minocycline may decrease BBB permeability, resulting in less perihematomal edema and decreased mass effect. Although numerous animal ICH models support minocycline's role as an inhibitor of MMP-9 and neuroprotectant, its use has never been studied in humans with ICH.

ELIGIBILITY:
Inclusion criteria:

1. Age 18-80 yo
2. Acute neurological deficit with corresponding ICH noted on head CT
3. Glasgow Coma Scale (GCS) > 8
4. Onset of symptoms within 12 hrs
5. < 30 ml of blood noted on initial CTH (30 ml hematoma volume is a noted independent marker between good and poor clinical outcome)
6. ICH score < 3
7. English/ Spanish speaking

Exclusion Criteria:

1. Allergy to tetracycline and tetracycline analogues
2. Pregnancy or suspected pregnancy
3. Hepatic and/or renal insufficiency (LFTs 3x greater than upper limit of normal; creatinine > 2 mg/dL)
4. Thrombocytopenia (plt count < 75,000)
5. History of intolerance to minocycline
6. Baseline modified Rankin score > 1
7. Stuporous or comatose (GCS < 8)
8. Presence of concomitant serious illness that would confound study, including serious psychiatric disease or prior suicide attempts.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06-27 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with Treatment-related Adverse Effects | day 90
  Treatment-related adverse effects as noted by package insert: fever, nausea, vomiting, C-diff, hepatic toxicity, dermatitis, anaphylaxis, renal injury)

SECONDARY OUTCOMES:
Volume (ml) of Perihematomal Edema | Change from baseline perihematomal edema volume to chronic (day 5-11) perihematomal edema volume
  Volumetric analysis (ml) computed from computed tomography head
modified Rankin score | day 90
  modified Rankin score (points ranging from 0 to 6)
Barthel Index | day 90
  Barthel Index score (points ranging from 0 to 100)
National Institutes of Health Stroke Scale Score | day 90
  National Institutes of Health Stroke Scale Score (points ranging from 0 to 42)
Glasgow Coma Score | day 90
  Glasgow Coma Score (points ranging from 3 to 15)

IPD SHARING:
Plan to Share IPD: No